CLINICAL TRIAL: NCT00273975
Title: A Randomised Open Label Multi-centre Trial to Evaluate the Pharmacokinetic, Efficacy and Safety Parameters of Nevirapine 150mg/m2 and Nevirapine 4 or 7 mg/kg When Administered in Combination With AZT and 3TC for 48 Weeks in Antiretroviral naïve Paediatric Patients.
Brief Title: Trial to Evaluate Steady State Pharmacokinetic Parameters, Efficacy and Safety of Nevirapine in Antiretroviral Drug naïve Pediatric Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1368
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Nevirapine
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
Trial to evaluate steady state pharmacokinetic parameters of nevirapine 150mg/m2 and nevirapine 4 or 7 mg/kg after 4 weeks, and efficacy and safety of the dosing when administered for 48 weeks in antiretroviral drug naïve paediatric patients.

DETAILED DESCRIPTION:
A randomised open label multi-centre trial to evaluate the pharmacokinetic, efficacy and safety parameters of nevirapine 150mg/m2 and nevirapine 4 or 7mg/kg when administered in combination with ZDV and 3TC for 48 weeks in antiretroviral naive pediatric patients.

Primary objective: To evaluate steady state pharmacokinetic parameters of nevirapine 150mg/m2 in antiretroviral drug naive pediatric patients.

Secondary objective: To assess efficacy and safety of nevirapine 150 mg/m2 and nevirapine 4/7mg/kg after 24 and 48 weeks of treatment

Study Hypothesis:

Evaluation of recent pharmacokinetic data has suggested that a dose based on body surface area rather than body weight might be a better therapeutic regimen to achieve steady state plasma concentrations. The goal in this study was to determine if a Nevirapine suspension dose of 150 mg/m2 BID, following a two week lead-in of 150 mg/m2 QD, produces plasma nevirapine steady state concentrations of 4 - 6 ?g/mL in all age groups as was observed in adult safety and efficacy trials.

Comparison(s):

ACTG 245

ELIGIBILITY:
Inclusion:

1. Male or female patients between 3 months and 16 years of age at day 28 of the study.
2. Evidence of HIV-1 infection
3. Patients who are antiretroviral drug naive
4. Plasma viral load detectable
5. CD4 >=50 cells/cc3
6. Written informed permission
7. Active assent given by the patient if the child is capable of understanding the given information
8. Reasonable probability for completion of the trial

Exclusion:

1. Any significant disease, other than HIV
2. Any acute illness within 2 weeks prior to Day 0
3. Patients requiring the continued use of inhibitors or inducers of P450 metabolic enzymes
4. Patients requiring systematic treatment with CYP3A4 substrates
5. Patients with malabsorption, severe chronic diarrhea
6. Receipt of any cytotoxic therapy for malignancy
7. Current grade 3 or 4 clinical or laboratory toxicity
8. Pregnancy or breast-feeding
9. Females of childbearing potential not using adequate contraception. allergy or known drug hypersensitivity to any of the study drugs intravenous drug abuse, alcohol or substance abuse

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 123
Dates: Start 2002-01; Primary Completion 2004-12 (Actual); Study Completion 2004-12

PRIMARY OUTCOMES:
Area under the concentration-time curve over one dosing interval (AUCτ) | 1, 3 and 6 hours on Day 28
Maximum observed concentration (Cmax) | 1, 3 and 6 hours on Day 28
Minimum observed concentration (Cmin) | 1, 3 and 6 hours on Day 28
Oral clearance (Dose/AUC) at steady state | 1, 3 and 6 hours on Day 28

SECONDARY OUTCOMES:
Change in HIV-1 RNA count | week 2, 4, 8, 12, 18, 24, 30, 36, 42,48
Virologic Response | 48 weeks
Time to Virologic Suppression | 48 weeks
Virologic Failure | 48 weeks
Time to Virologic Failure | 48 weeks
Treatment Failure | 48 weeks
Time to Treatment Failure | 48 weeks
Change in CD4+ cell count | week 2, 4, 8, 12, 18, 24, 30, 36, 42,48
Change in CD4+ percent | week 2, 4, 8, 12, 18, 24, 30, 36, 42,48
Occurrence of Adverse Events | 48 weeks
Occurrence of Rash | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. South Africa (Pty.) Ltd.
Locations (4):
- South Africa (4):
  - Groote Schuur Hospital, Cape Town
  - Boehringer Ingelheim Investigational Site, Pretoria
  - Boehringer Ingelheim Investigational Site, Soweto
  - Boehringer Ingelheim Investigational Site, Tygerberg